CLINICAL TRIAL: NCT00745004
Title: Ondansetron for the Treatment of IBS With Diarrhoea (IBS-D): Identifying the "Responder"
Brief Title: Ondansetron for the Treatment of IBS With Diarrhoea (IBS-D)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 08027
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2012-01

CONDITIONS: Irritable Bowel Syndrome With Diarrhoea
Keywords: IBS D
MeSH Terms: interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Ondansetron 4mg OD, dose titrated up to a maximum of 8mg tds or down to a minimum of 4mg alternate days.
  Interventions: Drug: Ondansetron
- 2 (Placebo Comparator): Placebo 1 capsule OD, dose titrated up to a maximum of 2 capsules tds or down to a minimum of 1 capsule alternate days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ondansetron — Over-encapsulated 4mg ondansetron tablets. Ondansetron 4mg OD, dose titrated up to a maximum of 8mg tds or down to a minimum of 4mg alternate days. For 5 weeks.
  Arms: 1
Drug: Placebo — Capsule matching over-encapsulated experimental drug. 1 capsule OD, dose titrated up to a maximum of 2 capsules tds or down to a minimum of 1 capsule alternate days. For 5 weeks.
  Arms: 2

SUMMARY:
Irritable bowel syndrome is a common condition affecting 1 in 10 of the population. About a third of these suffer from diarrhoea, which severely impairs their quality of life. Previous studies in Nottingham have suggested that some patients with diarrhoea may have an excess of a chemical called serotonin in their gut. Serotonin stimulates secretion and propulsion in the gut and contributes to diarrhoea. We are interested to see whether a drug, Ondansetron, which blocks the effect of serotonin, would improve symptoms in patients with IBS and diarrhoea. We think the drug may work better in people with a specific gene type so your genetic makeup may be of influence and we would like to test this. Because IBS symptoms fluctuate, one way to determine whether Ondansetron is effective is to perform a randomised placebo controlled trial in which neither the patient nor the doctor knows which medication is being taken in each part of the study.

ELIGIBILITY:
Inclusion Criteria:

* IBS-D patients meeting the Rome III criteria.
* Male or female aged 18-75 years
* Women of child bearing potential (who have a negative pregnancy test) must agree to use methods of medically acceptable forms of contraception during the study., (e.g. implants, injectables, combined oral contraceptives, sexual abstinence or vasectomised partners)
* Patients who are able to give informed consent.

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Patients that, in the opinion of the investigator, are considered unsuitable.
* Patients who have had abdominal surgery which may cause bowel symptoms similar to IBS (Please note, appendicectomy and cholecystectomy is not an exclusion)
* Patient unable to stop anti-diarrhoeal drugs
* Patients currently participating in another clinical trial or who have been in a trial in the previous three months

Since many patients will be on SSRIs or tricyclics antidepressants these will not be an exclusion criteria, provided they have been on medication at least 3 months and that the dose remains unaltered throughout the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the difference in average stool consistency during the last two week period of Ondansetron compared to placebo treatment. | 2 weeks

SECONDARY OUTCOMES:
1) Proportion of patients preferring ondansetron versus placebo 2) Proportion wanting to continue with ondansetron versus placebo 3) Difference between ondansetron and placebo periods. | Duration of study and post-study analysis

CONTACTS AND LOCATIONS:
Overall Officials: Robin Spiller, Principal Investigator — University of Nottingham; Peter Whorwell, MD, Principal Investigator — Manchester University NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - University Hospital of South Manchester NHS Foundation Trust, Manchester, Greater Manchester
  - University of Nottingham, Nottingham, Nottinghamshire

REFERENCES:
- [Derived] Tooth D, Garsed K, Singh G, Marciani L, Lam C, Fordham I, Fields A, Banwait R, Lingaya M, Layfield R, Hastings M, Whorwell P, Spiller R. Characterisation of faecal protease activity in irritable bowel syndrome with diarrhoea: origin and effect of gut transit. Gut. 2014 May;63(5):753-60. doi: 10.1136/gutjnl-2012-304042. Epub 2013 Aug 2. PMID 23911555